CLINICAL TRIAL: NCT01030822
Title: Booster Vaccination With Pneumococcal Vaccine GSK1024850A in Primed Children and Catch-up Vaccination in Unprimed Children
Brief Title: Booster and Catch-up Vaccination With Vaccine GSK1024850A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112909
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2017-01

CONDITIONS: Infections, Streptococcal
Keywords: Catch-up vaccination; Safety; Pneumococcal vaccine; Pneumococcal disease; Booster vaccination; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

ARMS (3):
- Group A (Experimental): Subjects previously primed with pneumococcal vaccine GSK1024850A in the first year of life and receiving a booster dose of GSK1024850A at 9-18 months of age.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A
- Group B (Experimental): Subjects previously primed with pneumococcal vaccine GSK1024850A in the first year of life and receiving a booster dose of GSK1024850A at 15-18 months of age.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A
- Group C (Experimental): Unprimed subjects receiving a catch-up vaccination (2+1 schedule) in the second year of life.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, administered as a single dose
  Arms: Group A; Group B
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, 3 doses
  Arms: Group C

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of a booster dose of pneumococcal vaccine GSK1024850A administered either at 9-18 months or 15-18 months of age in children primed in primary study NCT00814710.

This study also aims to assess the persistence of antibodies induced following primary vaccination with pneumococcal vaccine GSK1024850A in primary study NCT00814710 prior to booster vaccination and following vaccination in the present study at approximately 24 months of age.

The study is also designed to evaluate the immunogenicity, safety and reactogenicity of pneumococcal vaccine GSK1024850A when administered as a catch-up vaccination (2+1) in the second year of life in children unprimed with vaccine GSK1024850A in study NCT00814710.

DETAILED DESCRIPTION:
The study is randomized for primed subjects and non-randomized for unprimed subjects.

The protocol posting has been updated according to the amendment of the protocol dated 16 April 2010. The age range at the time of randomization of subjects primed in study NCT00814710 and the age range for booster vaccination of one of the groups has been extended.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects for whom the investigator believes that their parent(s)/ guardian(s) can and will comply with the requirements of the protocol.
* Written, signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child/ward. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

For primed subjects:

* Completion of the full vaccination course in study NCT00814710.
* 9-18 months of age at the time of randomization.
* Group A: 9-18 months of age at the time of booster vaccination.
* Group B: 15-18 months of age at the time of booster vaccination.

For unprimed subjects (Group C):

* Enrolled in study NCT00814710.
* 12-18 months of age at the time of first vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product within 30 days preceding the vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Administration of immunoglobulins and/or any blood products within three months preceding the vaccination or planned administration during the study period.
* Administration of any pneumococcal vaccine since the end of study NCT00814710.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2010-04-02; Primary Completion 2011-08-19 (Actual); Study Completion 2011-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- India (4):
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vellore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lalwani S. et al. Impact of age on booster responses to 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine in children in India. Abstract presented at the 6th Asian Congress of Pediatric Infectious Diseases (ACPID), Colombo, Sri Lanka, 28 Nov - 01 Dec 2012.
- [Derived] Lalwani S, Chatterjee S, Chhatwal J, Simon A, Ravula S, Francois N, Mehta S, Strezova A, Borys D. Randomized, open-label study of the impact of age on booster responses to the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in children in India. Clin Vaccine Immunol. 2014 Sep;21(9):1292-300. doi: 10.1128/CVI.00068-14. Epub 2014 Jul 9. PMID 25008901
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Synflorix 1 Group: Subjects who were previously primed with a 3-dose primary vaccination of Synflorix™ vaccine in the 10PN-PD-DIT-037 (111188) study, received a booster dose of Synflorix™ vaccine, administered intramuscularly in the right or left thigh, at 9-18 months of age.
- Synflorix 2 Group: Subjects who were previously primed with a 3-dose primary vaccination of Synflorix™ vaccine in the 10PN-PD-DIT-037 (111188) study, received a booster dose of Synflorix™ vaccine, administered intramuscularly in the right or left thigh, at 15-18 months of age.
- Tritanrix-HepB+Hiberix Group: Unprimed subjects who were previously vaccinated with Tritanrix™-HepB and Hiberix™ vaccines in the Control Group of the 10PN-PD-DIT-037 (111188) study, received a catch-up vaccination with Synflorix™ vaccine (2 primary doses +1 booster dose), administered intramuscularly in the right or left thigh, during their second year of life: 2+1 catch-up vaccination starting at 12-18 months of age with an interval of at least 8 weeks (56-118 days) between primary doses; the booster dose was administered at 18-24 months of age.
Period: Overall Study
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Started | 100 | 95 | 87
Completed | 69 | 71 | 61
Not Completed | 31 | 24 | 26
Not completed — Moved/migrated from study area | 6 | 7 | 3
Not completed — Withdrawal by Subject | 16 | 13 | 16
Not completed — Lost to Follow-up | 9 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group | Total
Number analyzed (Participants) | 100 | 95 | 87 | 282
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.5 (2.74) | 15.6 (1.27) | 16.1 (1.18) | 14.65 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 50 | 48 | 137
  Male | 61 | 45 | 39 | 145

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: Prior to booster vaccination (PRE), one month after booster vaccination (Month 1) and at approximately 24 months of age: at Month 15 for Synflorix 1 Group and at Month 9 for Synflorix 2 Group (24 months of age)
Population: The analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at the requested time points. Primary results are results one month after booster vaccination (Month 1).
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group
Number analyzed (Participants) | 89 | 71
µg/mL
  Anti-1 PRE: number analyzed (Participants) | 88 | 69
  Anti-1 PRE | 0.37 [0.29 to 0.48] | 0.31 [0.23 to 0.41]
  Anti-1 Month 1: number analyzed (Participants) | 80 | 61
  Anti-1 Month 1 | 4.78 [3.87 to 5.91] | 5.98 [4.54 to 7.9]
  Anti-1 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-1 24 months of age | 0.96 [0.68 to 1.37] | 1.37 [1 to 1.87]
  Anti-4 PRE: number analyzed (Participants) | 88 | 68
  Anti-4 PRE | 0.76 [0.58 to 1] | 0.58 [0.44 to 0.75]
  Anti-4 Month 1: number analyzed (Participants) | 81 | 63
  Anti-4 Month 1 | 7.28 [5.41 to 9.79] | 11.56 [7.96 to 16.79]
  Anti-4 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-4 24 months of age | 1.24 [0.9 to 1.7] | 2.29 [1.53 to 3.42]
  Anti-5 PRE: number analyzed (Participants) | 88 | 69
  Anti-5 PRE | 0.5 [0.4 to 0.63] | 0.38 [0.29 to 0.48]
  Anti-5 Month 1: number analyzed (Participants) | 81 | 62
  Anti-5 Month 1 | 5.86 [4.69 to 7.32] | 7.2 [5.25 to 9.86]
  Anti-5 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-5 24 months of age | 1.19 [0.86 to 1.65] | 2.03 [1.43 to 2.86]
  Anti-6B PRE: number analyzed (Participants) | 88 | 71
  Anti-6B PRE | 0.65 [0.5 to 0.85] | 0.49 [0.37 to 0.64]
  Anti-6B Month 1: number analyzed (Participants) | 81 | 64
  Anti-6B Month 1 | 2.82 [2.16 to 3.68] | 2.98 [2.05 to 4.32]
  Anti-6B 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-6B 24 months of age | 0.78 [0.54 to 1.11] | 0.9 [0.61 to 1.32]
  Anti-7F PRE: number analyzed (Participants) | 88 | 70
  Anti-7F PRE | 1.12 [0.92 to 1.38] | 0.93 [0.73 to 1.19]
  Anti-7F Month 1: number analyzed (Participants) | 81 | 63
  Anti-7F Month 1 | 6.3 [4.8 to 8.25] | 7.89 [5.91 to 10.54]
  Anti-7F 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-7F 24 months of age | 1.3 [0.96 to 1.76] | 1.98 [1.43 to 2.75]
  Anti-9V PRE: number analyzed (Participants) | 88 | 71
  Anti-9V PRE | 1.2 [0.94 to 1.52] | 0.96 [0.74 to 1.25]
  Anti-9V Month 1: number analyzed (Participants) | 81 | 64
  Anti-9V Month 1 | 8.03 [6.03 to 10.69] | 9.76 [7.08 to 13.44]
  Anti-9V 24 months of age: number analyzed (Participants) | 58 | 55
  Anti-9V 24 months of age | 1.7 [1.2 to 2.41] | 2.27 [1.64 to 3.14]
  Anti-14 PRE: number analyzed (Participants) | 89 | 70
  Anti-14 PRE | 1.76 [1.22 to 2.53] | 1.52 [1.08 to 2.15]
  Anti-14 Month 1: number analyzed (Participants) | 81 | 64
  Anti-14 Month 1 | 10.18 [7.6 to 13.65] | 11.85 [8.15 to 17.22]
  Anti-14 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-14 24 months of age | 3.02 [2.09 to 4.37] | 4.11 [2.98 to 5.67]
  Anti-18C PRE | 2.51 [1.94 to 3.23] | 1.55 [1.19 to 2.03]
  Anti-18C Month 1: number analyzed (Participants) | 81 | 63
  Anti-18C Month 1 | 33.39 [24.73 to 45.08] | 42.43 [31.48 to 57.2]
  Anti-18C 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-18C 24 months of age | 5.56 [3.84 to 8.05] | 10.04 [6.55 to 15.37]
  Anti-19F PRE: number analyzed (Participants) | 89 | 70
  Anti-19F PRE | 1.78 [1.34 to 2.36] | 1.23 [0.97 to 1.57]
  Anti-19F Month 1: number analyzed (Participants) | 81 | 64
  Anti-19F Month 1 | 13.68 [9.86 to 18.97] | 13.64 [9.42 to 19.76]
  Anti-19F 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-19F 24 months of age | 2.57 [1.81 to 3.65] | 4.15 [2.88 to 5.98]
  Anti-23F PRE: number analyzed (Participants) | 88 | 70
  Anti-23F PRE | 0.73 [0.55 to 0.97] | 0.65 [0.48 to 0.89]
  Anti-23F Month 1: number analyzed (Participants) | 81 | 63
  Anti-23F Month 1 | 5.54 [4.02 to 7.63] | 6.48 [4.69 to 8.96]
  Anti-23F 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-23F 24 months of age | 1.3 [0.88 to 1.91] | 1.38 [0.96 to 1.98]

2. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes
Description: as for outcome 1
Time Frame: Prior to vaccination (PRE), one month post-Dose 2 (Month 3), prior to (Month 6) and one month after the third (booster) vaccine dose (Month 7)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at the requested time points.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 81
µg/mL
  Anti-1 PRE | 0.04 [0.03 to 0.04]
  Anti-1 Month 3: number analyzed (Participants) | 69
  Anti-1 Month 3 | 2.5 [1.93 to 3.24]
  Anti-1 Month 6: number analyzed (Participants) | 65
  Anti-1 Month 6 | 1.03 [0.82 to 1.29]
  Anti-1 Month 7: number analyzed (Participants) | 54
  Anti-1 Month 7 | 3.32 [2.69 to 4.1]
  Anti-4 PRE: number analyzed (Participants) | 80
  Anti-4 PRE | 0.04 [0.03 to 0.05]
  Anti-4 Month 3: number analyzed (Participants) | 71
  Anti-4 Month 3 | 5.89 [4.23 to 8.22]
  Anti-4 Month 6: number analyzed (Participants) | 65
  Anti-4 Month 6 | 2.23 [1.85 to 2.69]
  Anti-4 Month 7: number analyzed (Participants) | 54
  Anti-4 Month 7 | 8.22 [5.92 to 11.42]
  Anti-5 PRE: number analyzed (Participants) | 80
  Anti-5 PRE | 0.05 [0.04 to 0.06]
  Anti-5 Month 3: number analyzed (Participants) | 71
  Anti-5 Month 3 | 2.81 [2.2 to 3.58]
  Anti-5 Month 6: number analyzed (Participants) | 65
  Anti-5 Month 6 | 1.39 [1.13 to 1.7]
  Anti-5 Month 7: number analyzed (Participants) | 54
  Anti-5 Month 7 | 5.32 [4.21 to 6.72]
  Anti-6B PRE: number analyzed (Participants) | 80
  Anti-6B PRE | 0.03 [0.03 to 0.04]
  Anti-6B Month 3: number analyzed (Participants) | 70
  Anti-6B Month 3 | 0.71 [0.53 to 0.95]
  Anti-6B Month 6: number analyzed (Participants) | 65
  Anti-6B Month 6 | 0.61 [0.47 to 0.78]
  Anti-6B Month 7: number analyzed (Participants) | 54
  Anti-6B Month 7 | 1.4 [1.04 to 1.88]
  Anti-7F PRE | 0.06 [0.05 to 0.08]
  Anti-7F Month 3: number analyzed (Participants) | 71
  Anti-7F Month 3 | 4.63 [3.38 to 6.34]
  Anti-7F Month 6: number analyzed (Participants) | 65
  Anti-7F Month 6 | 2.72 [2.28 to 3.24]
  Anti-7F Month 7: number analyzed (Participants) | 54
  Anti-7F Month 7 | 7.41 [5.87 to 9.34]
  Anti-9V PRE: number analyzed (Participants) | 80
  Anti-9V PRE | 0.04 [0.03 to 0.05]
  Anti-9V Month 3: number analyzed (Participants) | 71
  Anti-9V Month 3 | 2.09 [1.53 to 2.87]
  Anti-9V Month 6: number analyzed (Participants) | 65
  Anti-9V Month 6 | 1.74 [1.4 to 2.17]
  Anti-9V Month 7: number analyzed (Participants) | 54
  Anti-9V Month 7 | 4.88 [3.73 to 6.37]
  Anti-14 PRE: number analyzed (Participants) | 80
  Anti-14 PRE | 0.06 [0.05 to 0.08]
  Anti-14 Month 3: number analyzed (Participants) | 71
  Anti-14 Month 3 | 5.01 [3.75 to 6.69]
  Anti-14 Month 6: number analyzed (Participants) | 65
  Anti-14 Month 6 | 2.84 [2.25 to 3.57]
  Anti-14 Month 7: number analyzed (Participants) | 54
  Anti-14 Month 7 | 7.59 [5.87 to 9.8]
  Anti-18C PRE: number analyzed (Participants) | 80
  Anti-18C PRE | 0.04 [0.03 to 0.05]
  Anti-18C Month 3: number analyzed (Participants) | 70
  Anti-18C Month 3 | 29.1 [19.86 to 42.64]
  Anti-18C Month 6: number analyzed (Participants) | 65
  Anti-18C Month 6 | 12.44 [9.16 to 16.91]
  Anti-18C Month 7: number analyzed (Participants) | 54
  Anti-18C Month 7 | 75.19 [57.69 to 98.01]
  Anti-19F PRE: number analyzed (Participants) | 80
  Anti-19F PRE | 0.07 [0.05 to 0.1]
  Anti-19F Month 3: number analyzed (Participants) | 71
  Anti-19F Month 3 | 16.39 [11.15 to 24.1]
  Anti-19F Month 6: number analyzed (Participants) | 65
  Anti-19F Month 6 | 7.74 [5.85 to 10.24]
  Anti-19F Month 7: number analyzed (Participants) | 54
  Anti-19F Month 7 | 30.71 [23.76 to 39.68]
  Anti-23F PRE: number analyzed (Participants) | 80
  Anti-23F PRE | 0.04 [0.03 to 0.05]
  Anti-23F Month 3: number analyzed (Participants) | 71
  Anti-23F Month 3 | 1.13 [0.82 to 1.57]
  Anti-23F Month 6: number analyzed (Participants) | 65
  Anti-23F Month 6 | 0.85 [0.67 to 1.09]
  Anti-23F Month 7: number analyzed (Participants) | 54
  Anti-23F Month 7 | 2.15 [1.69 to 2.75]

3. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes (Persistence)
Description: as for outcome 1
Time Frame: Prior to booster vaccination (PRE) for the Synflorix 1 and Synflorix 2 Groups and prior to catch-up vaccination (PRE) for the Tritanrix-HepB+Hiberix Group
Population: The analysis was performed on the ATP cohort for persistence, which included all evaluable subjects for whom assay results for antibodies against at least one pneumococcal serotype were available before the administration of the booster dose of the Synflorix™ vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 89 | 90 | 84
µg/mL
  Anti-1: number analyzed (Participants) | 88 | 87 | 84
  Anti-1 | 0.37 [0.29 to 0.48] | 0.3 [0.24 to 0.39] | 0.04 [0.03 to 0.04]
  Anti-4: number analyzed (Participants) | 88 | 85 | 83
  Anti-4 | 0.76 [0.58 to 1] | 0.57 [0.45 to 0.72] | 0.04 [0.03 to 0.05]
  Anti-5: number analyzed (Participants) | 88 | 87 | 83
  Anti-5 | 0.5 [0.4 to 0.63] | 0.38 [0.31 to 0.47] | 0.05 [0.04 to 0.06]
  Anti-6B: number analyzed (Participants) | 88 | 90 | 83
  Anti-6B | 0.65 [0.5 to 0.85] | 0.51 [0.4 to 0.65] | 0.03 [0.03 to 0.04]
  Anti-7F: number analyzed (Participants) | 88 | 89 | 84
  Anti-7F | 1.12 [0.92 to 1.38] | 0.98 [0.79 to 1.23] | 0.06 [0.04 to 0.08]
  Anti-9V: number analyzed (Participants) | 88 | 90 | 83
  Anti-9V | 1.2 [0.94 to 1.52] | 0.98 [0.78 to 1.23] | 0.04 [0.03 to 0.05]
  Anti-14: number analyzed (Participants) | 89 | 89 | 83
  Anti-14 | 1.76 [1.22 to 2.53] | 1.37 [1 to 1.87] | 0.06 [0.05 to 0.08]
  Anti-18C: number analyzed (Participants) | 89 | 90 | 83
  Anti-18C | 2.51 [1.94 to 3.23] | 1.61 [1.26 to 2.05] | 0.04 [0.03 to 0.05]
  Anti-19F: number analyzed (Participants) | 89 | 88 | 83
  Anti-19F | 1.78 [1.34 to 2.36] | 1.36 [1.1 to 1.68] | 0.07 [0.05 to 0.09]
  Anti-23F: number analyzed (Participants) | 88 | 88 | 83
  Anti-23F | 0.73 [0.55 to 0.97] | 0.64 [0.49 to 0.85] | 0.04 [0.03 to 0.05]

4. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Persistence)
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: Prior to booster vaccination (PRE) for the Synflorix 1 and Synflorix 2 Groups and prior to catch-up vaccination (PRE) for the Tritanrix-HepB + Hiberix Group
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 87 | 84 | 78
Titer
  Opsono-1: number analyzed (Participants) | 87 | 84 | 77
  Opsono-1 | 16.5 [11.2 to 24.3] | 15.6 [10.5 to 23] | 4.4 [3.9 to 5]
  Opsono-4: number analyzed (Participants) | 85 | 81 | 67
  Opsono-4 | 70.3 [43.9 to 112.5] | 102.8 [66.4 to 159.1] | 6.2 [4.2 to 9.3]
  Opsono-5: number analyzed (Participants) | 87 | 81 | 78
  Opsono-5 | 11.9 [8.9 to 15.9] | 10.4 [7.8 to 13.7] | 4.2 [3.8 to 4.7]
  Opsono-6B: number analyzed (Participants) | 87 | 82 | 71
  Opsono-6B | 50.2 [30.7 to 82.1] | 62 [36.5 to 105.5] | 5.3 [3.9 to 7]
  Opsono-7F: number analyzed (Participants) | 87 | 84 | 65
  Opsono-7F | 1162.5 [910 to 1485] | 1551.1 [1269.4 to 1895.3] | 1186.4 [588.8 to 2390.7]
  Opsono-9V: number analyzed (Participants) | 83 | 82 | 60
  Opsono-9V | 430.4 [310.7 to 596.1] | 617.6 [477.6 to 798.6] | 192.6 [93.6 to 396.5]
  Opsono-14: number analyzed (Participants) | 85 | 79 | 69
  Opsono-14 | 206.4 [134.2 to 317.5] | 166.3 [105.7 to 261.6] | 13.5 [7.8 to 23.5]
  Opsono-18C: number analyzed (Participants) | 85 | 81 | 74
  Opsono-18C | 30.4 [20.7 to 44.6] | 23 [15.6 to 34] | 4.8 [3.8 to 6]
  Opsono-19F: number analyzed (Participants) | 86 | 82 | 76
  Opsono-19F | 43 [29.9 to 61.7] | 42.4 [29.5 to 60.8] | 4.2 [3.9 to 4.6]
  Opsono-23F: number analyzed (Participants) | 86 | 80 | 72
  Opsono-23F | 157 [83.2 to 296.3] | 531.1 [280.3 to 1006.4] | 41.9 [18.8 to 93.2]

5. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: as for outcome 4
Time Frame: Prior to booster vaccination (PRE), one month after booster vaccination (Month 1) and at approximately 24 months of age: at Month 15 for the Synflorix 1 Group and at Month 9 for Synflorix 2 Group (24 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 1 Group | Synflorix 2 Group
Number analyzed (Participants) | 87 | 65
Titer
  Opsono-1 PRE | 16.5 [11.2 to 24.3] | 14.3 [9.3 to 22.1]
  Opsono-1 Month 1: number analyzed (Participants) | 79 | 58
  Opsono-1 Month 1 | 1138.3 [828.6 to 1563.7] | 2096.7 [1464.8 to 3001.1]
  Opsono-1 24 months of age: number analyzed (Participants) | 57 | 54
  Opsono-1 24 months of age | 69.6 [40.1 to 121] | 173.8 [105.5 to 286.5]
  Opsono-4 PRE: number analyzed (Participants) | 85 | 63
  Opsono-4 PRE | 70.3 [43.9 to 112.5] | 101.6 [62.6 to 164.9]
  Opsono-4 Month 1: number analyzed (Participants) | 79 | 58
  Opsono-4 Month 1 | 3368.8 [2618 to 4334.9] | 7202.1 [5336.1 to 9720.6]
  Opsono-4 24 months of age: number analyzed (Participants) | 57 | 54
  Opsono-4 24 months of age | 557.4 [284 to 1093.9] | 2525.6 [1474.5 to 4325.9]
  Opsono-5 PRE: number analyzed (Participants) | 87 | 62
  Opsono-5 PRE | 11.9 [8.9 to 15.9] | 9.7 [7.2 to 13.1]
  Opsono-5 Month 1: number analyzed (Participants) | 79 | 58
  Opsono-5 Month 1 | 452.7 [353 to 580.6] | 834.6 [610.9 to 1140.2]
  Opsono-5 24 months of age: number analyzed (Participants) | 56 | 55
  Opsono-5 24 months of age | 45.7 [29.6 to 70.7] | 90.6 [54.8 to 149.8]
  Opsono-6B PRE: number analyzed (Participants) | 87 | 63
  Opsono-6B PRE | 50.2 [30.7 to 82.1] | 60 [32.9 to 109.3]
  Opsono-6B Month 1: number analyzed (Participants) | 79 | 57
  Opsono-6B Month 1 | 1556.6 [1090 to 2223] | 1781.2 [1042.5 to 3043.6]
  Opsono-6B 24 months of age: number analyzed (Participants) | 51 | 52
  Opsono-6B 24 months of age | 241.4 [127.7 to 456.4] | 287.5 [149 to 555]
  Opsono-7F PRE | 1162.5 [910 to 1485] | 1539.1 [1262.9 to 1875.6]
  Opsono-7F Month 1: number analyzed (Participants) | 79 | 57
  Opsono-7F Month 1 | 7814.8 [5984.8 to 10204.3] | 11064.4 [8182.9 to 14960.5]
  Opsono-7F 24 months of age: number analyzed (Participants) | 55 | 52
  Opsono-7F 24 months of age | 2891.2 [1954.4 to 4276.9] | 5371.9 [3712.4 to 7773.4]
  Opsono-9V PRE: number analyzed (Participants) | 83 | 63
  Opsono-9V PRE | 430.4 [310.7 to 596.1] | 704.9 [533.7 to 931.1]
  Opsono-9V Month 1: number analyzed (Participants) | 79 | 58
  Opsono-9V Month 1 | 4440 [3305.4 to 5964.2] | 7870.3 [5634.4 to 10993.4]
  Opsono-9V 24 months of age: number analyzed (Participants) | 49 | 52
  Opsono-9V 24 months of age | 1926.1 [1316.6 to 2817.9] | 3504.5 [2501 to 4910.6]
  Opsono-14 PRE: number analyzed (Participants) | 85 | 62
  Opsono-14 PRE | 206.4 [134.2 to 317.5] | 184 [109.8 to 308.2]
  Opsono-14 Month 1: number analyzed (Participants) | 79 | 57
  Opsono-14 Month 1 | 2057.1 [1569.6 to 2696.1] | 4407.5 [3193.2 to 6083.5]
  Opsono-14 24 months of age: number analyzed (Participants) | 56 | 53
  Opsono-14 24 months of age | 668.5 [403.1 to 1108.6] | 1641.2 [944.2 to 2852.9]
  Opsono-18C PRE: number analyzed (Participants) | 85 | 62
  Opsono-18C PRE | 30.4 [20.7 to 44.6] | 22.2 [14.1 to 35]
  Opsono-18C Month 1: number analyzed (Participants) | 79 | 58
  Opsono-18C Month 1 | 1889.7 [1429.4 to 2498.1] | 3643.2 [2572.2 to 5160.2]
  Opsono-18C 24 months of age: number analyzed (Participants) | 52 | 53
  Opsono-18C 24 months of age | 233.6 [142.2 to 383.8] | 1155 [662 to 2015]
  Opsono-19F PRE: number analyzed (Participants) | 86 | 63
  Opsono-19F PRE | 43 [29.9 to 61.7] | 34.7 [23.4 to 51.6]
  Opsono-19F Month 1: number analyzed (Participants) | 78 | 58
  Opsono-19F Month 1 | 1672.9 [1096.3 to 2552.7] | 2404.4 [1583.1 to 3651.6]
  Opsono-19F 24 months of age: number analyzed (Participants) | 51 | 53
  Opsono-19F 24 months of age | 107.3 [61.4 to 187.6] | 357.9 [218.9 to 585]
  Opsono-23F PRE: number analyzed (Participants) | 86 | 61
  Opsono-23F PRE | 157 [83.2 to 296.3] | 498.2 [231.4 to 1072.9]
  Opsono-23F Month 1: number analyzed (Participants) | 79 | 58
  Opsono-23F Month 1 | 3812.3 [2630.8 to 5524.5] | 5937.2 [3587.6 to 9825.5]
  Opsono-23F 24 months of age: number analyzed (Participants) | 54 | 55
  Opsono-23F 24 months of age | 1994.1 [959.7 to 4143.4] | 3018.5 [1389 to 6559.6]

6. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 75
Titer
  Opsono-1 PRE: number analyzed (Participants) | 74
  Opsono-1 PRE | 4.3 [3.9 to 4.8]
  Opsono-1 Month 3: number analyzed (Participants) | 68
  Opsono-1 Month 3 | 76.1 [49 to 118.2]
  Opsono-1 Month 6: number analyzed (Participants) | 64
  Opsono-1 Month 6 | 18.1 [11.5 to 28.4]
  Opsono-1 Month 7: number analyzed (Participants) | 54
  Opsono-1 Month 7 | 309.8 [203 to 472.9]
  Opsono-4 PRE: number analyzed (Participants) | 64
  Opsono-4 PRE | 5.8 [4 to 8.6]
  Opsono-4 Month 3: number analyzed (Participants) | 66
  Opsono-4 Month 3 | 2256.3 [1840 to 2766.8]
  Opsono-4 Month 6: number analyzed (Participants) | 63
  Opsono-4 Month 6 | 959.7 [727.2 to 1266.6]
  Opsono-4 Month 7: number analyzed (Participants) | 54
  Opsono-4 Month 7 | 2946.2 [2097.9 to 4137.4]
  Opsono-5 PRE | 4.2 [3.8 to 4.7]
  Opsono-5 Month 3: number analyzed (Participants) | 64
  Opsono-5 Month 3 | 76.3 [53.3 to 109.3]
  Opsono-5 Month 6: number analyzed (Participants) | 63
  Opsono-5 Month 6 | 24.6 [17 to 35.6]
  Opsono-5 Month 7: number analyzed (Participants) | 54
  Opsono-5 Month 7 | 212 [148.9 to 301.7]
  Opsono-6B PRE: number analyzed (Participants) | 68
  Opsono-6B PRE | 5.3 [3.9 to 7.2]
  Opsono-6B Month 3: number analyzed (Participants) | 63
  Opsono-6B Month 3 | 348.2 [165.7 to 731.6]
  Opsono-6B Month 6: number analyzed (Participants) | 61
  Opsono-6B Month 6 | 201.5 [98.2 to 413.5]
  Opsono-6B Month 7: number analyzed (Participants) | 53
  Opsono-6B Month 7 | 740.5 [419.6 to 1306.8]
  Opsono-7F PRE: number analyzed (Participants) | 63
  Opsono-7F PRE | 1106.8 [540.7 to 2265.9]
  Opsono-7F Month 3: number analyzed (Participants) | 67
  Opsono-7F Month 3 | 7462.5 [5653.9 to 9849.6]
  Opsono-7F Month 6: number analyzed (Participants) | 63
  Opsono-7F Month 6 | 6295.9 [4545 to 8721.4]
  Opsono-7F Month 7: number analyzed (Participants) | 54
  Opsono-7F Month 7 | 10104 [7377.8 to 13837.4]
  Opsono-9V PRE: number analyzed (Participants) | 58
  Opsono-9V PRE | 205.9 [98.7 to 429.4]
  Opsono-9V Month 3: number analyzed (Participants) | 61
  Opsono-9V Month 3 | 5792.5 [4586.3 to 7315.9]
  Opsono-9V Month 6: number analyzed (Participants) | 62
  Opsono-9V Month 6 | 3463.4 [2716.3 to 4416.1]
  Opsono-9V Month 7: number analyzed (Participants) | 53
  Opsono-9V Month 7 | 7000 [5265.1 to 9306.6]
  Opsono-14 PRE: number analyzed (Participants) | 67
  Opsono-14 PRE | 12.4 [7.1 to 21.6]
  Opsono-14 Month 3: number analyzed (Participants) | 65
  Opsono-14 Month 3 | 2359.8 [1576.1 to 3533.2]
  Opsono-14 Month 6: number analyzed (Participants) | 63
  Opsono-14 Month 6 | 1293.6 [886.8 to 1887.2]
  Opsono-14 Month 7: number analyzed (Participants) | 54
  Opsono-14 Month 7 | 3709.4 [2463.5 to 5585.2]
  Opsono-18C PRE: number analyzed (Participants) | 71
  Opsono-18C PRE | 4.8 [3.8 to 6.1]
  Opsono-18C Month 3: number analyzed (Participants) | 66
  Opsono-18C Month 3 | 2487.5 [1541.2 to 4014.8]
  Opsono-18C Month 6: number analyzed (Participants) | 62
  Opsono-18C Month 6 | 2546.4 [1755 to 3694.7]
  Opsono-18C Month 7: number analyzed (Participants) | 54
  Opsono-18C Month 7 | 8814.6 [6810.9 to 11407.7]
  Opsono-19F PRE: number analyzed (Participants) | 73
  Opsono-19F PRE | 4.2 [3.9 to 4.6]
  Opsono-19F Month 3: number analyzed (Participants) | 65
  Opsono-19F Month 3 | 1768.6 [1120.3 to 2792]
  Opsono-19F Month 6: number analyzed (Participants) | 62
  Opsono-19F Month 6 | 753.8 [497.3 to 1142.5]
  Opsono-19F Month 7: number analyzed (Participants) | 51
  Opsono-19F Month 7 | 3808.8 [2689.5 to 5393.9]
  Opsono-23F PRE: number analyzed (Participants) | 69
  Opsono-23F PRE | 38.7 [17.1 to 87.5]
  Opsono-23F Month 3: number analyzed (Participants) | 67
  Opsono-23F Month 3 | 3378.1 [2014.8 to 5664]
  Opsono-23F Month 6: number analyzed (Participants) | 62
  Opsono-23F Month 6 | 1868.2 [956.9 to 3647.5]
  Opsono-23F Month 7: number analyzed (Participants) | 53
  Opsono-23F Month 7 | 4357.3 [2246.9 to 8449.8]

7. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Persistence)
Description: Antibodies assessed for this outcome measure were those against cross-reactive pneumococcal serotypes 6A and 19A (ANTI-6A and -19A). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 89 | 89 | 84
µg/mL
  Anti-6A: number analyzed (Participants) | 89 | 87 | 83
  Anti-6A | 0.19 [0.14 to 0.26] | 0.22 [0.16 to 0.29] | 0.03 [0.03 to 0.04]
  Anti-19A: number analyzed (Participants) | 88 | 89 | 84
  Anti-19A | 0.31 [0.21 to 0.45] | 0.33 [0.25 to 0.45] | 0.06 [0.04 to 0.08]

8. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Antibodies assessed for this outcome measure were those against the cross-reactive pneumococcal serotypes 6A and 19A (ANTI-6A and -19A). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. Antibody concentrations < 0.05 µg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: Prior to booster vaccination (PRE), one month after booster vaccination (Month 1) and at approximately 24 months of age: at Month 15 for the Synflorix 1 Group and at Month 9 for the Synflorix 2 Group (24 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group
Number analyzed (Participants) | 89 | 70
µg/mL
  Anti-6A PRE | 0.19 [0.14 to 0.26] | 0.19 [0.14 to 0.27]
  Anti-6A Month 1: number analyzed (Participants) | 81 | 62
  Anti-6A Month 1 | 0.82 [0.59 to 1.14] | 0.95 [0.63 to 1.44]
  Anti-6A 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-6A 24 months of age | 0.32 [0.22 to 0.48] | 0.36 [0.22 to 0.59]
  Anti-19A PRE: number analyzed (Participants) | 88 | 70
  Anti-19A PRE | 0.31 [0.21 to 0.45] | 0.3 [0.22 to 0.41]
  Anti-19A Month 1: number analyzed (Participants) | 81 | 64
  Anti-19A Month 1 | 2.54 [1.61 to 4.03] | 2.87 [1.78 to 4.61]
  Anti-19A 24 months of age: number analyzed (Participants) | 59 | 55
  Anti-19A 24 months of age | 0.71 [0.45 to 1.14] | 1.33 [0.85 to 2.08]

9. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: as for outcome 7
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 81
µg/mL
  Anti-6A PRE: number analyzed (Participants) | 80
  Anti-6A PRE | 0.03 [0.03 to 0.04]
  Anti-6A Month 3: number analyzed (Participants) | 70
  Anti-6A Month 3 | 0.35 [0.25 to 0.5]
  Anti-6A Month 6: number analyzed (Participants) | 65
  Anti-6A Month 6 | 0.33 [0.24 to 0.45]
  Anti-6A Month 7: number analyzed (Participants) | 54
  Anti-6A Month 7 | 0.76 [0.53 to 1.09]
  Anti-19A PRE | 0.06 [0.04 to 0.08]
  Anti-19A Month 3: number analyzed (Participants) | 71
  Anti-19A Month 3 | 2.49 [1.77 to 3.51]
  Anti-19A Month 6: number analyzed (Participants) | 65
  Anti-19A Month 6 | 1.94 [1.44 to 2.61]
  Anti-19A Month 7: number analyzed (Participants) | 54
  Anti-19A Month 7 | 7.91 [5.62 to 11.13]

10. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Persistence)
Description: OPA titers against cross-reactive pneumococcal serotypes 6A and 19A (Opsono-6A and -19A) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 86 | 82 | 78
Titer
  Opsono-6A: number analyzed (Participants) | 86 | 82 | 72
  Opsono-6A | 21.1 [13.2 to 33.6] | 30.1 [18.4 to 49.3] | 10.3 [6.3 to 17]
  Opsono-19A | 9.7 [6.8 to 13.7] | 7.4 [5.7 to 9.7] | 4.8 [4 to 5.7]

11. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: as for outcome 10
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix 1 Group | Synflorix 2 Group
Number analyzed (Participants) | 86 | 63
Titer
  Opsono-6A PRE | 21.1 [13.2 to 33.6] | 27.1 [15.7 to 47]
  Opsono-6A Month 1: number analyzed (Participants) | 79 | 57
  Opsono-6A Month 1 | 168.7 [96.3 to 295.5] | 262.5 [135.4 to 509]
  Opsono-6A 24 months of age: number analyzed (Participants) | 54 | 53
  Opsono-6A 24 months of age | 62.2 [33.7 to 114.8] | 96.6 [45.4 to 205.6]
  Opsono-19A PRE | 9.7 [6.8 to 13.7] | 7 [5.3 to 9.3]
  Opsono-19A Month 1: number analyzed (Participants) | 78 | 57
  Opsono-19A Month 1 | 161.6 [93.7 to 278.5] | 385.6 [223.4 to 665.5]
  Opsono-19A 24 months of age: number analyzed (Participants) | 53 | 51
  Opsono-19A 24 months of age | 17.8 [9.8 to 32.1] | 60 [33 to 109.2]

12. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: as for outcome 10
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 75
Titer
  Opsono-6A PRE: number analyzed (Participants) | 69
  Opsono-6A PRE | 10.2 [6.1 to 17.1]
  Opsono-6A Month 3: number analyzed (Participants) | 65
  Opsono-6A Month 3 | 324.9 [176.1 to 599.5]
  Opsono-6A Month 6: number analyzed (Participants) | 63
  Opsono-6A Month 6 | 329 [181 to 598.2]
  Opsono-6A Month 7: number analyzed (Participants) | 52
  Opsono-6A Month 7 | 616.2 [369.2 to 1028.5]
  Opsono-19A PRE | 4.8 [4 to 5.8]
  Opsono-19A Month 3: number analyzed (Participants) | 64
  Opsono-19A Month 3 | 506.6 [305.5 to 840.1]
  Opsono-19A Month 6: number analyzed (Participants) | 61
  Opsono-19A Month 6 | 402.1 [248.9 to 649.5]
  Opsono-19A Month 7: number analyzed (Participants) | 54
  Opsono-19A Month 7 | 1770.9 [1190.6 to 2634]

13. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) (Persistence)
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 100 EL.U/mL. Antibody concentrations < 100 EL.U/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 89 | 90 | 82
EL.U/mL | 776.3 [629 to 958.2] | 618.6 [488.2 to 783.9] | 71.6 [62.3 to 82.2]

14. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: as for outcome 13
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group
Number analyzed (Participants) | 89 | 71
EL.U/mL
  Anti-PD PRE | 776.3 [629 to 958.2] | 654.7 [497.9 to 860.9]
  Anti-PD Month 1: number analyzed (Participants) | 89 | 61
  Anti-PD Month 1 | 3704.2 [2825.6 to 4856] | 5297.6 [3934 to 7133.8]
  Anti-PD 24 months of age: number analyzed (Participants) | 59 | 54
  Anti-PD 24 months of age | 1337.3 [953.8 to 1875] | 2191.9 [1582.5 to 3036]

15. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: as for outcome 13
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 79
EL.U/mL
  Anti-PD PRE | 72.5 [62.9 to 83.7]
  Anti-PD Month 3: number analyzed (Participants) | 70
  Anti-PD Month 3 | 527.7 [397.4 to 700.9]
  Anti-PD Month 6: number analyzed (Participants) | 65
  Anti-PD Month 6 | 443.2 [333.1 to 589.6]
  Anti-PD Month 7: number analyzed (Participants) | 54
  Anti-PD Month 7 | 1727.2 [1306.6 to 2283.3]

16. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: Within the 4-day follow-up period (Days 0-3) after the booster dose for the Synflorix 1 and Synflorix 2 Groups and across doses for the Tritanrix-HepB + Hiberix Group
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine dose administration documented and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 93 | 85 | 82
Participants
  Any Pain | 31 | 25 | 26
  Grade 3 Pain | 2 | 4 | 5
  Any Redness | 16 | 12 | 11
  Grade 3 Redness | 2 | 0 | 1
  Any Swelling | 14 | 14 | 16
  Grade 3 Swelling | 4 | 1 | 2

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness (Irr./Fuss.), Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]),. Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal everyday activities. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal everyday activities. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 92 | 85 | 82
Participants
  Any Drowsiness | 5 | 4 | 5
  Grade 3 Drowsiness | 0 | 0 | 2
  Related Drowsiness | 4 | 4 | 3
  Any Fever | 20 | 13 | 22
  Grade 3 Fever | 0 | 1 | 0
  Related Fever | 19 | 13 | 21
  Any Irr./Fuss. | 19 | 9 | 12
  Grade 3 Irr./Fuss. | 1 | 1 | 1
  Related Irr./Fuss. | 15 | 9 | 9
  Any Loss of Appetite | 14 | 9 | 10
  Grade 3 Loss of Appetite | 0 | 2 | 0
  Related Loss of Appetite | 9 | 8 | 9

18. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31-day follow-up period (Days 0-30) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 100 | 95 | 87
Participants | 7 | 1 | 5

19. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life- threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity.
Time Frame: After the first vaccination up to study end (from Month 0 to Month 15)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Number analyzed (Participants) | 100 | 95 | 87
Participants | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 4 days post-vaccination; Unsolicited AEs: during the 31 days post-vaccination after booster dose in the Synflorix 1 and Synflorix 2 Groups and across doses in the Tritanrix-HepB+Hiberix Group; SAEs: from Month 0 to Month 15.
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Tritanrix-HepB+Hiberix Group
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/95 | 1/87
Other Adverse Events (participants affected / at risk) | 48/100 | 29/95 | 38/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix 1 Group (N=100) | Synflorix 2 Group (N=95) | Tritanrix-HepB+Hiberix Group (N=87)
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix 1 Group (N=100) | Synflorix 2 Group (N=95) | Tritanrix-HepB+Hiberix Group (N=87)
Pain (General disorders) | 31/93 | 25/85 | 26/82
Redness (General disorders) | 16/93 | 12/85 | 11/82
Swelling (General disorders) | 14/93 | 14/85 | 16/82
Drowsiness (General disorders) | 5/92 | 4/85 | 5/82
Fever (≥38°C) (General disorders) | 20/92 | 13/85 | 22/82
Irritability (General disorders) | 19/92 | 9/85 | 12/82
Loss of appetite (General disorders) | 14/92 | 9/85 | 10/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.